CLINICAL TRIAL: NCT02580214
Title: A Protocol Of Perioperative Care Plus Immunonutrition Enhances Recovery After Total Hip Arthroplasty. A Randomized Pilot Study
Brief Title: Immunonutrition in Total Hip Arthroplasty
Acronym: Immunehip
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of Mato Grosso (Other)
Responsible Party: Principal Investigator, Jose Eduardo de Aguilar-Nascimento, Chair Professor, MD, PhD, Federal University of Mato Grosso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FUMatogrossoSul
Record Dates: First submitted 2015-10-15; First posted 2015-10-20 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Arthroplasty, Hip Replacement; Perioperative Care; Nutritional Support

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acerto (Experimental): Preoperative immune nutrition for 5 days (Impact, Nestle) Preoperative fasting of 2h with a drink containing 12% maltodextrine No intravenous fluids postoperatively
  Interventions: Dietary Supplement: Impact
- Control (No Intervention): No immune nutrition Preoperative fasting of 6-8 h Crystalloid intravenous fluids until PO day 1

INTERVENTIONS:
Dietary Supplement: Impact — 600 ml of Impact, Nestle for 5 days prior to surgery
  Arms: Acerto

SUMMARY:
The aim of this pilot study was to investigate whether the use of a multimodal protocol of preoperative care plus preoperative immune nutrition would decrease the length of stay and acute phase inflammation in patients submitted to total hip arthroplasty (THA). The study was designed to be randomized and controlled, but not double blind. The patients were randomized to receive either preoperative care based on evidence plus immune nutrition for 5 days prior to surgery (Acerto group) or traditional preoperative care (control group). Main endpoints were length of stay and acute-phase postoperative response

DETAILED DESCRIPTION:
A large broad of evidence has shown that traditional perioperative care have a weak scientific basis and needs to be changed. Multimodal or fast-track protocols of perioperative care for abdominal surgery have been associated with lower morbidity, lower costs and faster postoperative recovery when compared to traditional care . Similarly the prescription of perioperative immune nutrition for 5-7 days before major abdominal surgery may decrease the risk of infections and reduce postoperative length of stay (LOS). Interestingly there is lack of studies on multimodal protocols of enhanced recovery and on immune nutrition in elective total hip arthroplasty (THA). In Brazil, the ACERTO (an acronym in Portuguese for acceleration of postoperative recovery) protocol is a multimodal protocol of perioperative care that includes: shortening of preoperative fasting with carbohydrates (CHO)-rich drinks up to 2h before surgery, restriction of intravenous fluids and early postoperative re-feeding and mobilization. Recently as a dynamic protocol the Acerto protocol included the recommendation of perioperative immune nutrition. All the elements of the protocol are based on evidence and are recommended by various international guidelines and consensus. Thus, the aim of this pilot study was to investigate whether the use of the Acerto multimodal protocol plus preoperative immune nutrition would decrease the length of stay and acute phase inflammation in patients submitted to THA.

METHODS This was a prospective randomized pilot study. All procedures were performed at São Mateus Hospital (Cuiabá, Brazil) from May 2012 to February 2013. The study was approved by the Research Ethics Committee of the Júlio Müller University Hospital (Federal University of Mato Grosso) and all patients signed a term of informed consent.

Inclusion and exclusion criteria. The investigators included adult patients of both sex having a hip osteoarthrosis and candidates of elective THA. Patients were excluded if they had fasting glycemia greater than 200mg/dl; acquired immunodeficiency (AIDS); renal failure (creatinin above 2 mg/dl); cirrhosis; moderate or serious Alzheimer's disease (clinical dementia rating score between 2 and 3); an American Society of Anesthesiologists (ASA) score higher than 2; previous spinal surgery (arthrodesis) or THA (reviewing or changing the prosthetic); and severe malnutrition (history of loss of 10% of body weight over the last 6 months). The investigators also excluded patients who did not have their blood samples taken at the scheduled time and those who broke perioperative protocol, e.g. the non-intake of the immune supplement in the Acerto group.

Design of the study. Patients were consecutively included and randomized into two groups: Group Control and ACERTO group with the aid of electronic software of random numbers available at www.graphpad.com. All patients were assessed by a multidisciplinary team, who carried out a nutrition assessment, preoperative education, and collected the relevant anthropometric, biochemical and clinical data.

Anesthesia and operative technique. Antibiotic prophylaxis was done with 2g of intravenous kefazolin at the time of anesthetic induction. Measures were taken against postoperative nausea and vomiting (PONV) according to the protocol applied by the anesthesia team and will be discussed in this paper. Preoperative sedation was done with intravenous midazolam (0.03 to 0.1mg/kg) and propofol (30 to 60 mcg/kg/min) No general anesthetic was applied in both groups. All subjects received epidural neuro-axis blockage at L3-L4 space with ropivacain 7.5% to 10% (150-200mg) and morphine chlorate 2mg (30 to 50 micrograms/kg). The surgical access of the hip was done by anterior-lateral approach. The investigators used in all cases hybrid type total arthroplasty (cementation of the femoral component and fixation of the acetabular component by means of pressure fitting of the implant to the bone and the addition of screws to the acetabular cup when necessary).

Carbohydrate drink Patients belonging to the Acerto group received a drink (200 mL) containing water plus 12% maltodextrin 2h before the induction of anesthesia.

Immune supplementation therapy. The patients in the ACERTO group received an immune supplement containing arginine, w-3 fatty acids, nucleotides, and vitamins (Impact; Nestlé; Sao Paulo, Brazil. Formula: proteins: 23% (77% calcium caseinate, 23% arginine); carbohydrates: 52% (100% maltodextrin); lipids: 25% (68% fish oil; 20% medium-chain triglycerides and 12% corn oil), vitamins and electrolytes) for five days prior to surgery, with a daily dosage of thress units (600ml per day in total).

Blood samples. Blood samples were collected preoperatively and at the 2nd PO day and assayed for CRP assay.

Criteria for hospital discharge.

Discharge was signed by an orthopedic surgeon if all of these five parameters were fulfilled:

1. patient is confident and willing to go home,
2. no pain or pain controlled by oral analgesics,
3. walking alone or with minimal help,
4. no fever or signs of postoperative infection, and
5. accepting normal oral diet

Outcome variables The main outcome variable was the postoperative length of stay. As secondary outcome variables it was compared the evolution of serum C-reactive protein (CRP) overtime.

Statistical analysis. The calculation of the sample was based on the premise that the intervention with the Acerto Project protocol would reduce the hospital stay length by 50%. For a β error (type II) of 20% and an α error (type I) of 5%, it was calculated that 15 patients in each group would be sufficient for this study. Investigators used paired and unpaired t-test when samples were homogeneous or the Mann-Whitney test or the Wilcoxon test if samples were heterogeneous. Categorical variables were compared by the chi square test or Fisher exact test. Statistical analyses were made using the Minitab 14 and the null hypothesis rejection was fixed at 0.05 (α=5%).

ELIGIBILITY:
Inclusion Criteria:

* We included adult patients (18-80 y/o) of both sex having a hip osteoarthrosis and candidates of elective THA.

Exclusion Criteria:

* Patients were excluded if they had fasting glycemia greater than 200mg/dl
* Acquired immunodeficiency (AIDS)
* Renal failure (creatinin above 2 mg/dl)
* Cirrhosis
* Moderate or serious Alzheimer's disease (clinical dementia rating score between 2 and 3)
* An American Society of Anesthesiologists (ASA) score higher than 2
* Previous spinal surgery (arthrodesis) or THA (reviewing or changing the prosthetic)
* Severe malnutrition (history of loss of 10% of body weight over the last 6 months).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-05; Primary Completion 2014-03 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Length of postoperative stay | up to 30 days of the postoperative course
  days of postoperative stay until discharge up to 30 days

SECONDARY OUTCOMES:
Serum C-reactive protein | preoperative and 2nd PO day
  Blood samples collected at anesthesia induction and again at PO day 2 to C-reactive protein assay

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroclinica, Cuiabá, Mato Grosso, Brazil

REFERENCES:
- [Derived] Alito MA, de Aguilar-Nascimento JE. Multimodal perioperative care plus immunonutrition versus traditional care in total hip arthroplasty: a randomized pilot study. Nutr J. 2016 Apr 2;15:34. doi: 10.1186/s12937-016-0153-1. PMID 27038614